CLINICAL TRIAL: NCT07071090
Title: An Open-Label Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, and Preliminary Efficacy of DC50292A Tablet in Patients With MTAP-deleted Advanced or Metastatic Solid Tumors
Brief Title: A Study of DC50292A Tablet in Patients With MTAP-deleted Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Heronova Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHRC-CRDC05-01-01
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor Malignancies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DC50292A (Experimental): All enrolled subjects will receive DC50292A orally. Doses will be escalated from low to high：40 mg, 100 mg, 200 mg, 400 mg, 600 mg, 900 mg.
  Interventions: Drug: DC50292A

INTERVENTIONS:
Drug: DC50292A — DC50292A tablet

SUMMARY:
This study employs a non-randomized, open-label design to evaluate the safety, tolerability, pharmacokinetic (PK) profile, and preliminary efficacy of DC50292A tablets in patients with MTAP-deficient advanced or metastatic solid tumors. The study consists of two parts: dose escalation and dose expansion.

DETAILED DESCRIPTION:
Dose Escalation Phase: The dose escalation study will first be conducted using an accelerated titration "3+3" design, progressing from lower to higher dose levels. Six dose groups are planned: 40 mg, 100 mg, 200 mg, 400 mg, 600 mg, and 900 mg (subject to adjustment based on study results, such as adding intermediate dose levels). The 40 mg group will follow an accelerated titration design, enrolling 1-6 subjects, while the 100-900 mg groups will enroll 3-6 subjects per cohort.

Each dose group will undergo: Single-dose administration (C0D1-C0D5): A single dose on C0D1, followed by PK blood sampling from C0D2 to C0D5.

Cycle 1 (C1D1-C1D21): Starting from C1D1 (after C0D5), subjects will receive daily dosing for 3 weeks, followed by a 3-day break (until C1D25 pre-dose) for dose-limiting toxicity (DLT) assessment, along with PK and pharmacodynamic (PD) sample collection and analysis. Subsequent cycles (C2D1-CnD28): Continuous dosing in subsequent cycles, with adjustments and optimizations based on cumulative safety, PK, and PD data. If no DLT-based stopping criteria are met during the observation period, the dose will escalate to the next level. After the DLT observation period, eligible subjects may continue treatment with DC50292A until disease progression, intolerable toxicity, initiation of new antitumor therapy, withdrawal of consent, voluntary discontinuation, death, loss to follow-up, or other protocol-specified termination criteria-whichever occurs first. Dose Expansion Phase: after determining the maximum tolerated dose (MTD) in the escalation phase, two optimal doses (≤MTD) will be selected for expansion based on cumulative efficacy, safety, and PK data. Each expansion cohort will enroll 8 subjects, receiving oral DC50292A in an optimized regimen (tentatively once daily in 4-week cycles) until meeting discontinuation criteria (as above).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signs the informed consent form, demonstrates understanding of the study, and is willing and able to comply with all trial procedures.
2. Age ≥18 years, regardless of gender.
3. Patients with histologically and/or cytologically confirmed solid tumors who are assessed by the investigator as having locally advanced, recurrent, or metastatic disease and have failed standard treatments at the current stage.
4. At least one measurable lesion as per RECIST v1.1 criteria, assessed via imaging (tumor lesions located in previously irradiated areas or those having undergone other local-regional therapies are generally not considered measurable unless clear progression is confirmed by the investigator).
5. MTAP deficiency, defined by one of the following: willingness to provide sufficient archived tumor tissue or fresh biopsy samples for MTAP testing; or documentation of MTAP homozygous deletion via NGS/IHC or loss of MTAP protein expression in tissue; or availability of a prior NGS report (within 3 years) confirming MTAP homozygous deletion or an IHC report confirming loss of MTAP expression, as accepted by the investigator.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
7. Life expectancy ≥3 months.
8. Absence of severe hematological, hepatic, renal, coagulation, or cardiac dysfunction.
9. Male and female participants of childbearing potential must agree to use effective contraception from the time of signing the informed consent form until 3 months after the last dose of the study drug. Female participants of childbearing potential must have a negative serum pregnancy test result prior to the first dose of the study medication.

Exclusion Criteria:

1. Received chemotherapy, radiotherapy, biologics, endocrine therapy, immunotherapy, or other antitumor treatments within 4 weeks or 5 half-lives (whichever is shorter) before the first dose of the study drug, including: nitrosoureas or mitomycin C within 6 weeks prior; oral fluoropyrimidines or small-molecule targeted agents within 2 weeks or 5 half-lives (whichever is shorter); Chinese herbal medicines with antitumor indications within 2 weeks prior.
2. Received any non-marketed investigational drugs or therapies within 4 weeks prior to the first dose.
3. Undergone major organ surgery (excluding needle biopsy or surgery for pathologic fractures), significant trauma, or planned elective surgery during the trial within 4 weeks prior.
4. Used CYP3A4-sensitive substrates, strong inhibitors/inducers, CYP2C8-sensitive substrates, or P-gp inhibitors (see Appendix 3) within 14 days or 5 half-lives (whichever is shorter) prior.
5. Previously treated with PRMT5 or MAT2A inhibitors.
6. QTc interval ≥480 ms (mean of 3 measurements) on screening/baseline 12-lead ECG.
7. Prior allogeneic hematopoietic stem cell/bone marrow transplantation or solid organ transplantation, or current use of immunosuppressants/anti-rejection drugs.
8. Known allergy to any active/inactive ingredient of the study drug.
9. Adverse reactions from prior antitumor therapy not resolved to CTCAE v5.0 Grade ≤1 (except non-risks like alopecia, Grade 2 peripheral neuropathy, or stable hypothyroidism on hormone replacement).
10. Hepatitis B (HBsAg+ with HBV-DNA ≥2500 copies/mL or 500 IU/mL), HCV (HCV-RNA > lower limit of detection), HIV-positive, or syphilis (both specific/non-specific antibodies positive).
11. Symptomatic/active CNS metastases, leptomeningeal disease, or spinal cord compression. Asymptomatic CNS metastases may enroll if:

    1. Measurable extracranial lesions per RECIST v1.1;
    2. No new/progressive CNS lesions for ≥4 weeks with stable neurologic symptoms;
    3. No seizures/increased intracranial pressure;
    4. No steroids/antiepileptics/dehydrants for ≥2 weeks.
12. Clinically significant third-space fluid accumulation (e.g., massive ascites/pleural effusion).
13. Cardiovascular Disease: severe arrhythmias (e.g., ventricular arrhythmias requiring intervention, AV block II-III); ACS, CHF, aortic dissection, stroke, or Grade ≥3 cardiovascular events within 6 months; NYHA Class ≥II or high-risk structural heart disease; uncontrolled hypertension (SBP ≥150 mmHg and/or DBP ≥95 mmHg); QTc prolongation risks (e.g., heart failure, uncorrected hypokalemia, congenital/family history of long QT syndrome, concomitant QT-prolonging drugs).
14. Systemic treatment for active infection within 4 weeks prior.
15. Acute esophageal/GI diseases affecting drug absorption (e.g., bowel obstruction, Crohn's disease, ulcerative colitis, short bowel syndrome).
16. Pulmonary Disease: interstitial lung disease (ILD), pulmonary fibrosis, or drug-induced pneumonitis requiring treatment.
17. Other Severe Conditions: hepatic, renal, neurologic/psychiatric, endocrine, hematologic, or immune disorders compromising study participation.
18. Other malignancies within 5 years (except cured malignancies like basal/ squamous cell skin cancer, low-risk prostate cancer, papillary thyroid cancer, or excised in situ cancers).
19. Known alcohol/drug dependence.
20. Psychiatric disorders or poor adherence.
21. Pregnant or breastfeeding women.
22. Investigator's Discretion: any other clinical/laboratory abnormalities deemed unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | 12 months
  Incidence and severity of adverse events as assessed by CTCAE Version 5.0

SECONDARY OUTCOMES:
PK profile of DC50292A | From time zero up to 96 hours post-dose
  Peak Concentration (Cmax): The maximum plasma concentration of the drug.
PK profile of DC50292A | From time zero up to 96 hours post-dose
  Area Under the Curve from Time Zero to the Last Measurable Concentration (AUC0-t): The area under the plasma concentration-time curve from time zero to the last measurable concentration.
PK profile of DC50292A | From time zero up to 96 hours post-dose
  Area Under the Curve from Time Zero Extrapolated to Infinity (AUC0-∞): The area under the plasma concentration-time curve from time zero extrapolated to infinity.
PK profile of DC50292A | From time zero up to 96 hours post-dose
  Time to Reach Peak Concentration (Tmax): The time at which the peak plasma concentration is reached.
PK profile of DC50292A | From time zero up to 96 hours post-dose
  Elimination Half-Life (T1/2): The time required for the plasma concentration to decrease by half.
Overall response rate (ORR) | Up to 12 months
  Overall response rate (ORR) based on RECIST v1.1 as assessed by the investigator
Progression-free Survival (PFS) | Up to 12 months
  Progression-free survival (PFS) based on RECIST v1.1 as assessed by the investigator

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shandong Cancer Hospital, Jinan, Shandong
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No